CLINICAL TRIAL: NCT02820311
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Positive-Controlled, 4-Period Crossover Thorough QT Study to Evaluate the Effect of a Single Dose of TD-4208 on Cardiac Repolarization in Healthy Subjects
Brief Title: Thorough QT (TQT) Study of TD-4208 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mylan Inc. (Industry)
Collaborators: Theravance Biopharma (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0136
Record Dates: First submitted 2016-06-23; First posted 2016-06-30 (Estimated); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Cardiac Repolarization in Healthy Subjects
Keywords: Thorough QT (TQT); cardiac safety
MeSH Terms: interventions — revefenacin; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- TD-4208 175 mcg (Experimental): double-blind
  Interventions: Drug: TD-4208 175 mcg
- TD-4208 700 mcg (Experimental): double-blind
  Interventions: Drug: TD-4208 700 mcg
- Placebo for TD-4208 (Placebo Comparator): double-blind
  Interventions: Drug: Placebo for TD-4208
- Moxifloxacin 400 mg (Active Comparator): open-label
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: TD-4208 175 mcg — via nebulizer
  Other Names: revefenacin
  Arms: TD-4208 175 mcg
Drug: TD-4208 700 mcg — via nebulizer
  Other Names: revefenacin
  Arms: TD-4208 700 mcg
Drug: Placebo for TD-4208 — via nebulizer
  Arms: Placebo for TD-4208
Drug: Moxifloxacin 400 mg — oral
  Other Names: Avelox
  Arms: Moxifloxacin 400 mg

SUMMARY:
The purpose of this study is to evaluate if TD-4208, an investigational drug being developed to treat people with chronic obstructive pulmonary disease (COPD), has any effect on the electrical activity of the heart.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index (BMI) of 19 to 32 kg/m2, inclusive, and weight of at least 55 kg.
* Subject is able to communicate well with the investigator and to comply with the study procedures, requirements, and restrictions.

Exclusion Criteria:

* Subject has a prior history of myocardial infarction, acute coronary syndrome, cerebrovascular accident, transient ischemic attack, ventricular tachycardia, atrial fibrillation, personal or known family history of congenital long QT syndrome or known family history of sudden death with unknown cause, a pacemaker or implantable cardioverter defibrillator, cardiac or cerebral stent placement or angioplasty, or clinically significant valvular heart disease.
* Subject has evidence or history of clinically significant allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematologic, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurological disease.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Change-from-baseline in corrected QT | Predose to 24 hours postdose

SECONDARY OUTCOMES:
Maximum Plasma Concentration Cmax | Predose to 24 hours postdose
Adverse Events | Predose to 24 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Theravance Biopharma
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No